CLINICAL TRIAL: NCT03331224
Title: Endoscopic Treatment of Non-variceal Upper GI-bleeding With High Risk of Recurrency - OTSC (Over-the-scope-clip) Versus Standard Therapy (STING2)
Acronym: STING2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Collaborators: University Hospital Freiburg (Other); University Hospital Ulm (Other); University Hospital Goettingen (Other); Evangelisches Krankenhaus Düsseldorf (Other); University Hospital, Essen (Other); University of Leipzig (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STING2
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Acute Upper Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTSC (Experimental): Initial treatment with the OTSC for non-variceal upper GI-bleedings with high risk of recurrency.
  Interventions: Device: OTSC
- Standard therapy (Active Comparator): Endoscopic standard therapy (two techniques e.g. clip and injection)
  Interventions: Device: Endoscopic Standard therapy (combining two methods)

INTERVENTIONS:
Device: OTSC — OTSC placement
  Arms: OTSC
Device: Endoscopic Standard therapy (combining two methods) — endoscopic standard therapy (two methods, e.g. clip and injection)
  Arms: Standard therapy

SUMMARY:
Prospective-randomized multi-center trial. Patients with high risk of recurrent GI-bleeding (non-variceal) are identified and randomized into either endoscopic treatment with the OTSC [Over The Scope Clip] or endoscopic standard therapy. Hypothesis: Endoscopic therapy with OTSC is superior to standard therapy regarding technical success and rebleeding.

DETAILED DESCRIPTION:
Prospective-randomized multi-center trial. Patients with high risk of recurrent GI-bleeding (non-variceal) are identified (Rockall Score > 6) and randomized into either endoscopic treatment with the OTSC [Over The Scope Clip] or endoscopic standard therapy. 100 Patients are planned. Hypothesis: Endoscopic therapy with OTSC is superior to standard therapy regarding technical success and rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* upper GI-bleeding (non-variceal) with high risk of recurrency
* 18 years and older

Exclusion Criteria:

* variceal-bleeding
* under 18 years
* pregnancy or nursing period
* malignancy
* need for surgical treatment (for example perforation with peritonitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Persistent bleeding or Rebleeding with 7 days | 7 days

SECONDARY OUTCOMES:
blood units transfused | 30 days
duration of hospital stay | 30 days
duration of intensive care unit stay | 30 days
30 d Mortality | 30 days
Amount of endoscopic reinterventions | 7 days
Necessity of surgical or angiographic therapy | 7 days
Complications during or after OTSC (Over The Scope Clip) placement | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meier B, Wannhoff A, Denzer U, Stathopoulos P, Schumacher B, Albers D, Hoffmeister A, Feisthammel J, Walter B, Meining A, Wedi E, Zachaus M, Pickartz T, Kullmer A, Schmidt A, Caca K. Over-the-scope-clips versus standard treatment in high-risk patients with acute non-variceal upper gastrointestinal bleeding: a randomised controlled trial (STING-2). Gut. 2022 Jul;71(7):1251-1258. doi: 10.1136/gutjnl-2021-325300. Epub 2022 Mar 23. PMID 35321938